CLINICAL TRIAL: NCT06544395
Title: Efficacy of Non-invasive Neuromodulation Treatments for Post-COVID-19 Sequelae in Patients With Musculoskeletal, Respiratory and Neurological Conditions Due to Impaired Taste and Smell.
Brief Title: Efficacy of Non-invasive Neuromodulation Treatments for COVID-19 Sequelae
Acronym: COVID-19
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Gema Leon (Other)
Responsible Party: Principal Investigator, GEMA LEÓN BRAVO, Principal Investigator, Clinica Gema Leon
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: NO INVASIV NEUROMOD COVID-19; NO INVASIVE NEUROM-COVID-19 (Other: CLINICA DE FISIOTERAPIA GEMA LEÓN)
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Covid-19 Recurrent
Keywords: Covid-19; Non Invasive Neuromodulation; Smell
MeSH Terms: conditions — COVID-19; Anosmia | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients receiving non invasive neuromodulation treatment. (Experimental): Patients without previous pathology of any kind who have passed the Covid19 and have respiratory, neurological or musculoskeletal sequelae; who will receive non invasive neuromodulation treatment.
  Interventions: Device: Non invasive neuromodulation therapy
- Patients receiving traditional treatment. (Active Comparator): Patients receiving only traditional therapy. Patients without previous pathology of any kind who have passed the Covid19 and have respiratory, neurological or musculoskeletal sequelae; who will receive treatment of traditional therapy.
  Interventions: Other: Manual therapy
- Patients receiving placebo treatment. (Placebo Comparator): Patients receiving placebo. Patients without previous pathology of any kind who have passed the Covid19 and have respiratory, neurological or musculoskeletal sequelae; to those who will be administered placebo (device off, without emitting).
  Interventions: Device: Placebo with non invasive neuromodulation

INTERVENTIONS:
Device: Non invasive neuromodulation therapy — In the 4 studies, the intervention consisted of 15 sessions spread over 5 weeks.
  Each intervention lasted 60 minutes. The intensity will be programmed in all sessions at Low, following the Arndt-Schulz law. The treatment was distributed in 3 phases: phase 1 of preparation, phase 2 to reduce fatigue and phase 3 to enhance autonomic improvement.
  Arms: Patients receiving non invasive neuromodulation treatment.
Other: Manual therapy — Common manual therapy administered for said pathology by traditional physiotherapy and therapeutic exercise.
  Arms: Patients receiving traditional treatment.
Device: Placebo with non invasive neuromodulation — In the 4 studies, the intervention consisted of 15 sessions spread over 5 weeks.
  Each intervention lasted 60 minutes. The treatment was carried out with the machine turned off.
  Arms: Patients receiving placebo treatment.

SUMMARY:
The goal of this clinical trial is to demonstrate the effectiveness of non-invasive Neuromodulation as a therapy in neurological, respiratory and musculoskeletal pathologies derived from the consequences of Covid-19. It will also estimate the impact of non-invasive neuromodulation treatment on the functionality and quality of life of patients with COVID-19 sequelae.The main question it aim to answer is:

- Is non-invasive neuromodulation effective as a therapy in neurological, respiratory and musculoskeletal pathologies derived from the consequences of Covid-19.

Researchers will compare non-invasive neuromodulation to a placebo (treatment with the machine turned off).

Participants will:

* Be evaluated before starting treatment.
* Be evaluated 3 weeks after.
* Be evaluated at 5 weeks, or 15 sessions or completion of treatment.
* Be evaluated 6 weeks after finishing the treatment or 11 weeks after starting treatment.

DETAILED DESCRIPTION:
The waves of Sars-Cov-2 disease continue to be continuous and we are increasingly aware of the consequences it causes both in the respiratory system, musculoskeletal system and in the central and peripheral nervous system.

Likewise, non-invasive neuromodulation acts with a pump of ions, generating endogenous stimuli that modulate the central nervous system.

The aim of this clinical trial is to demonstrate the effectiveness of non-invasive Neuromodulation as a therapy in neurological, respiratory and musculoskeletal pathologies derived from the consequences of Covid-19.

To carry out this study, pain was measured with the visual analogue scale. It was also measured the joint amplitude, a muscle assessment with the help of a strength dynamometer, the patient's independence with the Katz index and the functionality of the lower or upper limbs, depending on the affected joint.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 60.
* Patients with a positive diagnosis of COVID-19.
* Patients with post-COVID-19 sequelae with musculoskeletal, respiratory or neurological symptoms due to taste or smell lasting at least 30 days, with no history of respiratory and/or neurological and/or musculoskeletal diseases.
* Patients who signed the informed consent.

Exclusion criteria:

* Patients aged before 18 years and after 60 years.
* Healthy people with no history of neurological, neurological and/or respiratory and/or musculoskeletal diseases
* Patients with secondary diseases that could directly affect the systems to be evaluated who were not diagnosed positive for COVID-19.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
ad hoc patient survey | one month
  survey of patients about conditions diagnosed during the illness and those they suffer from after infection that are directly related to abnormalities to be assessed.
sex, age, vaccination and number of months with symptoms | one month
  Nominal variables such as sex, age, vaccination and number of months with symptoms
Number of participants with musculoskeletal, respiratory and neurological sequelae of taste and smell after COVID-19 | three months

SECONDARY OUTCOMES:
SDOQ-NS questionnaire for social impairments due to loss of smell | two months
  Assess the quality of life impairments of patients with olfactory dysfunction. In a scale of 0 to 3, with higher scores reflecting better olfactory-specific
SF12 Quality of Life Questionnaire | two months
  Assesses the impact of health on an individual's everyday life. Scores above 50 indicate a better-than-average health-related quality of life, while scores below 50 suggest below-average health.
Brief Smell Identification Test: Assessment of smell. | two months
  Assesses the ability to recognize familiar odors. A 12-item questionnaire. For each item, a microcapsule containing a familiar odor is scratched with a pencil and placed under the participant's nose.
  The total score is the number of odors that are correctly recognized. Missing responses are assigned a partial score of 0.25. If more than 2 responses are missing, the entire test is treated as missing.
EuroQoL 5-D scale (validated translation into Spanish) for quality of life. | two months
  Quality of life related to health.
  Questionaire with two parts:
  1. Descriptive system (5 items). Minimum value: 1 (absence of dificulties). Maximum value: 3 (plenty of difficulties). Optimal value: 1.
  2. Visual analogical scale (EVA). Minimum value: 0 (worst imaginable state of health). Maximum value: 100 (best imaginable state of health). Optimal value: 100.
upper limb functional index | two months
  It is used to evaluate functional impairment in people with upper extremity musculoskeletal dysfunction. 25 questions assessing the level of difficulty in performing activities of daily living using your upper extremities, including household and work activities, hobbies, lifting a bag of food, washing your scalp, pushing on your hands, driving, etc. Patients respond to each item by circling the number that best describes their level of difficulty.
lower limb functional index | two months
  Valid patient-rated outcome measure to measure lower extremity function. The lower the score the greater the disability. The minimal detectable change is 9 scale points.
Visual analogue scale (VAS), for pain assessment | two months
  Intensity of pain. Minimum value: 0 (absence of pain). Maximum value: 10 (unbearable pain). Optimal value: 0.
Sensory assessment for pain and light touch | two months
  The sensory exam involves evaluation of pain and light touch. Test pain using a sharp object. At minimum, test the shoulders, arms and legs, comparing side to side and proximal to distal areas. In any area where the patient complains of sensory loss or hypersensitivity, more detailed testing may be required.
  For light touch, uses your fingertips or a wisp of cotton, lightly stroke the skin and determine if the patient feels this symmetrically in all areas tested. At minimum, test the shoulders, arms and legs, comparing side to side and proximal to distal areas.
Sadoul's dyspnea rating scale. | two months
  Respiratory evaluation. Minimum value: 0 (absence of dyspnea). Maximum value: 5 (dyspnea occurs with minimal efforts). Optimal value: 0.
measurement of lung function with spirometry and lung volume testing | three months
  measurement of lung function with spirometry and lung volume testing (measurement of maximum inspiratory and expiratory pressures (Pimax and Pemax, respectively)

CONTACTS AND LOCATIONS:
Overall Officials: GEMA LEÓN BRAVO, Principal Investigator — Departamento de Enfermería, Farmacología y Fisioterapia de la Universidad de Córdoba
Locations (1):
- Gema León Physiotherapy and Rehabilitation Clinic, Córdoba, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No